CLINICAL TRIAL: NCT03478046
Title: Alterations in Phosphorylated Fetuin-A, a Novel Regulator of Insulin Action in Insulin Resistance and Metabolic Syndrome: Effects of Lifestyle Modification
Brief Title: Fetuin-A Phosphorylation Status in Insulin Resistance and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Suresh Mathews, Associate Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-210-MR0710
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese individuals (Experimental): Apparently healthy, weight-stable, obese and physically inactive male volunteers will be recruited. Intervention is an 8 to 10% weight loss induced by chronic exercise training and dietary modification
  Interventions: Other: Weight loss

INTERVENTIONS:
Other: Weight loss — Compare the total and temporal changes in fetuin-A phosphorylation and insulin resistance that occur with an 8 to 10% weight loss induced by chronic exercise training and dietary modification

SUMMARY:
Fetuin-A has been identified as a novel physiological regulator of insulin action in vitro, in intact cells and in vivo in animals. Previous research has shown that circulating levels of fetuin-A were increased in animal models of insulin resistance and diabetes. Additionally, several human investigation studies demonstrate a correlation of fetuin-A levels with body mass index, insulin resistance, and a fatty liver. Recently, the investigators have elucidated the role of fetuin-A phosphorylation in the regulation of insulin action, demonstrating that phosphorylation is critical for the inhibitory activity of fetuin-A. The objectives of this study are twofold: (1) Quantitate phosphorylated fetuin-A levels in individuals with insulin resistance and metabolic syndrome, and (2) Investigate the effects of lifestyle modifications (acute or chronic exercise and dietary modifications) on fetuin-A phosphorylation and insulin sensitivity.

DETAILED DESCRIPTION:
There are several objectives of this study: (1) Quantitate phosphorylated fetuin-A levels and the daily variation in these levels in individuals with insulin resistance and metabolic syndrome; (2) Investigate the short-term responses of fetuin-A phosphorylation and changes in insulin resistance that occur with a single session of aerobic exercise; (3) Characterize and compare the total and temporal changes in fetuin-A phosphorylation and insulin resistance that occur with an 8 to 10% weight loss induced by chronic exercise training and dietary modification, and; (4) Investigate the influence of weight loss on the short-term responses of fetuin-A phosphorylation and changes in insulin resistance that occur with a single session of aerobic exercise. Our hypothesis is that phosphofetuin-A levels are tightly correlated with insulin resistance and that lifestyle modifications will improve insulin sensitivity and decrease phosphorylated fetuin-A levels.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 65 years of age
* obese (BMI > 30 kg⋅m2 or % fat > 30, and waist girth > 88 cm)
* weight stable over the previous 6 months

Exclusion Criteria:

* smoker
* documented cardiovascular or metabolic disease
* currently taking medication to alter lipid or glucose metabolism
* practicing regular leisure physical activity over the previous 6 months
* engaged in strenuous vocational activity over the previous 6 months
* signs or symptoms of latent heart disease
* conditions that would preclude treadmill walking

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10-10 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Total plasma fetuin-A and phosphorylated fetuin-A | Total fetuin-A and phosphorylated fetuin-A levels will be measured once every 4 weeks until participant achieves a targeted weight-loss goal of 8-10%. It is anticipated that most participants will achieve their weight-loss goal within 6-10 months.
  Measure total fetuin-A and phosphorylated fetuin-A levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Mathews, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ren G, Bowers RL, Kim T, Mahurin AJ, Grandjean PW, Mathews ST. Serum fetuin-A and Ser312 phosphorylated fetuin-A responses and markers of insulin sensitivity after a single bout of moderate intensity exercise. Physiol Rep. 2021 Mar;9(5):e14773. doi: 10.14814/phy2.14773. PMID 33650781